CLINICAL TRIAL: NCT02944994
Title: Effectiveness of a Unified Transdiagnostic Treatment in Routine Clinical Care
Brief Title: Effectiveness of a Unified Transdiagnostic Treatment in Routine Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H-33257; K23MH103396 (NIH)
Record Dates: First submitted 2016-04-08; First posted 2016-10-26 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Anxiety; Traumatic Stress Disorders; Depression
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Traumatic; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unified Protocol (Experimental): Unified Protocol-psychotherapy
  Interventions: Other: Unified protocol
- Routine Care (Experimental): Routine Care psychotherapy comparison
  Interventions: Other: Routine Care

INTERVENTIONS:
Other: Unified protocol — This is a transdiagnostic cognitive behavioral therapy
  Arms: Unified Protocol
Other: Routine Care — This arm will reflect typical care received in routine mental health care
  Arms: Routine Care

SUMMARY:
The purpose of this study is to examine effectiveness and implementation for the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in trauma exposed veterans.

DETAILED DESCRIPTION:
Anxiety and mood diagnoses are chronic and devastating with respect to costs to the individual and the healthcare system, and are more prevalent than any other class of disorders. When these disorders present concurrently, the significant public health implications and societal costs are intensified. Despite high rates of comorbidity and underlying mechanistic similarities between treatment protocols, single disorder evidence- based psychotherapy protocols for these disorders have traditionally been recommended to treat emotional disorders sequentially. Moreover, when clinicians are presented with complex case presentations, they are often unprepared to treat them and move away from evidence-based approaches, potentially increasing the burden on the mental health system. The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders (UP) is an innovative transdiagnostic protocol with promising evidence for successful treatment of emotional disorders, both for standalone and comorbid presentations, including the classification of not otherwise specified (NOS) disorders. To date, there have only been efficacy trials of the UP, which limit generalizability and do not address the larger public health impact and effectiveness in routine clinical care settings with both psychiatric and medical comorbidity. To address this critical limitation, the applicant proposes a pilot feasibility, acceptability, and tolerability study of the UP in patients with diverse psychiatric and medical comorbidity to manualized supportive therapy within a hospital. The deployment focused model (DFM) will inform design and statistical analyses. An additional aim includes determining the feasibility, acceptability, perceived fit and satisfaction of the UP in clinic settings through surveying and interviewing stakeholders in the system that are implementing the UP through the study. Consultation with stakeholders can minimize the time required to collect and assess fit within the larger system and, therefore, minimizes the time lag between science and practice in routine care settings. This study addresses an important public health concern by examining the effectiveness of the UP in a new population as a strategy for treatment of common and debilitating mental disorders in routine care settings. Furthermore, the proposed research aims will complement a comprehensive training plan to prepare the applicant to become an independent investigator with expertise in implementation science and effectiveness research. Results from the study will provide important information about whether or not this efficacious treatment can be effective, efficient, and ready for implementation in routine care settings in which psychiatric and medical comorbidity are common. This study will also serve as a model of deploying efficacious treatments into generalist clinics.

ELIGIBILITY:
Inclusion Criteria for Veteran Participants:

* VA Boston Health Care Patient:

Definition: Currently enrolled as a patient at VA Boston Healthcare System

* Diagnosis of an emotional disorder Definition: Diagnostic and Statistical Manual-5 (DSM-5) diagnosis of any emotional disorder (anxiety disorder, traumatic stress disorders, or unipolar depression)
* Cognitive Functioning:

Definition: free of cognitive impairment demonstrated by ability to understand and provide consent

* Psychotherapy:

Definition: not currently in psychotherapy for an emotional disorder treated in the study

Stakeholder Inclusion Criteria

* Provider Status:

Definition: Providing or overseeing mental health treatment in VA Boston Healthcare System and VA Puget Sound Healthcare System

Exclusion Criteria:

* Veteran Participant Exclusionary Criteria
* Current diagnosis of substance dependence (but not abuse)
* Primary diagnosis of bipolar disorder
* Current diagnosis of psychosis
* High suicidal risk (plan with intent)
* Recent change in psychiatric medications (< 3 months prior to entering the study).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-12; Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
Barriers and facilitators that impact implementation of the intervention measured by the Consolidated Framework for Implementation Research (CFIR) | One time assessment, occurring on 1 day, approximately 4 months after treatment initiation
  These interviews will occur at one time point and will be analyzed with Qualitative Comparative Analyses guided by the Consolidated Framework for Implementation Research. Qualitative analyses are often descriptive in nature and a summary of common themes are reported to speak to factors impacting implementation of the intervention in this population. NVivo software will be used to aggregate the qualitative interviews from all participants and highlight the common themes across CFIR interviews
Change in clinician administered Anxiety Disorders Interview Scheduled will be used to generate clinical diagnoses for mental health disorders | 7 months
  Change will be examined from baseline through the end of treatment. For each participant it will be reported if there was a change in each participants clinician administered diagnostic assessment and the resulting clinician severity rating for each mental health diagnosis. This assessment will be used in conjunction with the CAPS-5 (outcome 3) to inform the presence or absence of clinical diagnoses at baseline and follow-up. Each has it's own metric, but can be used to show the presence or absence of a clinical level of the diagnosis
Change in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) will be used to asses the presence or absence of a clinical diagnosis of PTSD | 7 months
  Change will be examined from baseline through the end of treatment. For each participant it will be reported if there was a change in each participants clinician administered diagnostic assessment and the resulting severity rating for a PTSD diagnosis. This assessment will be used in conjunction with the ADIS-5 (outcome 2) to inform the presence or absence of clinical diagnoses at baseline and follow-up. Each has it's own metric, but can be used to show the presence or absence of a clinical level of the diagnosis. They cannot be combine into one variable unless a dichotomous score is calculated to indicate a clinical diagnosis more broadly is present versus absent.

CONTACTS AND LOCATIONS:
Overall Officials: Cassidy Gutner, PhD, Principal Investigator — Boston University
Locations (1):
- VA Boston Healthcare System, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gutner CA, Song J, Canale CA, Suvak MK, Litwack SD, Niles BL, Stirman SW. A pilot randomized effectiveness trial of the unified protocol in trauma-exposed veterans. Depress Anxiety. 2022 Dec;39(12):813-823. doi: 10.1002/da.23288. Epub 2022 Oct 18. PMID 36258655